CLINICAL TRIAL: NCT02288520
Title: Therapeutic Strategy in Rheumatology When Faced With a Patient Treated With Methotrexate (MTX) for Rheumatoid Arthritis (RA).
Brief Title: Therapeutic Strategy in Patients Treated With Methotrexate for Rheumatoid Arthritis
Acronym: STRATEGE
Status: Completed | Type: Observational
Sponsor: Nordic Pharma SAS (Industry)
Responsible Party: Sponsor
Other Study IDs: STRATEGE
Record Dates: First submitted 2014-11-07; First posted 2014-11-11 (Estimated); Last update posted 2016-06-02 (Estimated); Status verified 2015-10

CONDITIONS: Rheumatoid Arthritis
Keywords: Methotrexate; Therapeutic strategy
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a longitudinal, observational, prospective, multicentre study conducted in metropolitan France, among a representative sample of office-based or mixed practice rheumatology doctors.

The aim of this study is to describe in real life, the therapy strategy when faced with a patient treated with methotrexate as a monotherapy consulting for rheumatoid arthritis and the impact on the progression of the disease at 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient, ambulatory, seen in a rheumatology consultation.
* With a confirmed diagnosis of RA (ACR 1987 or ACR/EULAR 2010 criteria) receiving a disease-modifying treatment with methotrexate as a monotherapy.
* With clinical, functional, structural and/or therapeutic disease progression, for whom the rheumatologist intends to change the therapeutic treatment of the RA .
* Informed about the computer processing of their medical data and their right of access and correction.

Exclusion Criteria:

* Patient not treated with methotrexate for their RA.
* Already treated with a biotherapy or receiving other synthetic DMARDs (disease-modifying antirheumatic drugs) in combination with methotrexate .
* Participating in a clinical trial in rheumatology.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Rheumatoid arthritis (RA) patients with clinical, functional, structural and/or therapeutic disease progression, for whom the rheumatologist intends to change the therapeutic treatment of the RA will be asked to participate from RA treatment change (inclusion visit) up to 6 months after inclusion.
Sampling Method: Non-Probability Sample
Enrollment: 854 (Actual)
Dates: Start 2014-09; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Therapeutic options and Impact on the progression of the disease (EULAR (European League Against Rheumatism) criteria (change in DAS28 (Disease Activity Score 28) | Patients are included at the time of the change in the treatment of the RA and followed up to 6 months
  The distribution of the various therapeutic options will be described overall. Their impact on the progression of the RA will be assessed at 6 months according to the EULAR (European League Against Rheumatism) criteria (change in DAS28 (Disease Activity Score 28) score during the study)

SECONDARY OUTCOMES:
Patient's satisfaction using a 4-point verbal scale | 6 months after inclusion
  Satisfaction will be assessed using a 4-point verbal scale.
Medical economic aspect (cost/benefit ratio) | 6 months after inclusion
  The cost/benefit ratio of each therapeutic strategy will be described.

CONTACTS AND LOCATIONS:
Overall Officials: Hélène HERMAN DEMARS, MD, Study Director — Nordic Pharma
Locations (1):
- Nordic Pharma, Paris, France

REFERENCES:
- [Derived] Gaujoux-Viala C, Hudry C, Zinovieva E, Herman-Demars H, Flipo RM. MTX optimization or adding bDMARD equally improve disease activity in rheumatoid arthritis: results from the prospective study STRATEGE. Rheumatology (Oxford). 2021 Dec 24;61(1):270-280. doi: 10.1093/rheumatology/keab274. PMID 33774669